CLINICAL TRIAL: NCT04823507
Title: Photobiomodulation for Concussions: the Use of the ImPACT® Test to Assess Improvement in Cognition and Symptomatology
Brief Title: Photobiomodulation for Concussions: the Use of the ImPACT® Test as an Assessment Tool
Status: Completed | Type: Observational
Sponsor: Meditech Rehabilitation Centre (Other)
Responsible Party: Sponsor
Other Study IDs: BFX1
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Concussion, Photobiomodulation, ImPACT
MeSH Terms: conditions — Brain Concussion; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Concussion patients treated with Photobiomodulation: * Patients between the ages of 15-65 years clinically diagnosed with a mild Traumatic Brain Injury by a health professional and currently not undergoing any treatment during a 1 year period from January 2018 to December 2018.
  * Documentation of the history of a qualifying mild Traumatic Brain Injury within 3 months of traumatic incident and/or diagnosis with persistent symptomatology after 3 months. For reference, International Classification of Diseases, Tenth Revision (ICD-10) clinical criteria require a history of TBI and the presence of three or more of the following eight symptoms: 1) headache, 2) dizziness, 3) fatigue, 4) irritability, 5) insomnia, 6) concentration or 7) memory difficulty, and 8) intolerance of stress, emotion, or alcohol4.
  Interventions: Device: BIOFLEX DUO+

INTERVENTIONS:
Device: BIOFLEX DUO+ — * Data scores will be collected for patients who initially underwent the Workplace Post-Injury 1 test of the ImPACT® test system prior to PBM treatment.
  * Patients were treated with photobiomodulation using the BIOFLEX® DUO+ system that utilized a 180 bulb Light Emitting Diode (LED) array followed by laser probes. Both delivery methods were applied to the cervical spine and the cranium, and both entailed the use of red light at 660 nm wavelength and near-infrared light at 830-840 nm wavelength. Treatment is provided three times per week on alternating days with weekends off for 4 weeks for a total of 12 treatments utilizing Health Canada approved device specific protocol guidelines for treatment of the cervical spine.
  * Data scores will be collected for a second ImPACT® test using the Workplace Post-Injury 2 test.
  * Results of the Post-Injury 1 test and the Post-Injury 2 test will be compared.
  Other Names: ImPACT test

SUMMARY:
Brain photobiomodulation (PBM) therapy is an innovative modality for the stimulation of neural activity in order to improve brain function and is currently under investigation as a treatment for several diverse neurological disorders. Our emphasis on this study is to review the use of PBM as a treatment modality for concussions and the use of ImPACT® (Immediate Post-Concussion Assessment and Cognitive Testing) test to assess improvement in cognition and symptomatology in patients with post-concussion syndrome (PCS) treated with PBM.

DETAILED DESCRIPTION:
* This will be a retrospective, single arm, unmasked, clinical study.
* Data scores will be collected for patients who initially underwent the Workplace Post-Injury 1 test of the ImPACT® test system prior to PBM treatment.
* Patients were treated with photobiomodulation using the BIOFLEX® DUO+ system that utilized a 180 bulb Light Emitting Diode (LED) array followed by laser probes. Both delivery methods were applied to the cervical spine and the cranium, and both entailed the use of red light at 660 nm wavelength and near-infrared light at 830-840 nm wavelength. Treatment is provided three times per week on alternating days with weekends off for 4 weeks for a total of 12 treatments utilizing Health Canada approved device specific protocol guidelines for treatment of the cervical spine.
* Data scores will be collected for a second ImPACT® test using the Workplace Post-Injury 2 test.
* Results of the Post-Injury 1 test and the Post-Injury 2 test will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 15-65 years clinically diagnosed with a mild Traumatic Brain Injury by a health professional and currently not undergoing any treatment during a 1 year period from January 2018 to December 2018.
* Documentation of the history of a qualifying mild Traumatic Brain Injury within 3 months of traumatic incident and/or diagnosis with persistent symptomatology after 3 months. For reference, International Classification of Diseases, Tenth Revision (ICD-10) clinical criteria require a history of TBI and the presence of three or more of the following eight symptoms: 1) headache, 2) dizziness, 3) fatigue, 4) irritability, 5) insomnia, 6) concentration or 7) memory difficulty, and 8) intolerance of stress, emotion, or alcohol4.

Exclusion Criteria:

* Any positive findings on imaging studies
* A diagnosis of or a family history of neuropsychiatric co-morbidity.
* Any additional diagnoses compounding the diagnosis of a concussion or mild traumatic brain injury (TBI)
* Currently undergoing any type of therapy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected for all patients diagnosed with post-concussion syndrome who sought consult and treated using photobiomodulation therapy at Meditech Rehabilitation Centre using the BIOFLEX® DUO+ system
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Improvement in ImPACT test scores after treatment with Photobiomodulation. | 4 weeks
  • Statistically significant change in measured metrics for Workplace Post injury 2 ImPACT® outcome scores compared to Workplace Post injury 1 ImPACT® scores for patients in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zitney, MD, Principal Investigator — Meditech Rehabilitation Centre
Locations (1):
- Meditech Rehabilitation Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only overall outcomes will be shared.

REFERENCES:
- [Background] Salehpour F, Mahmoudi J, Kamari F, Sadigh-Eteghad S, Rasta SH, Hamblin MR. Brain Photobiomodulation Therapy: a Narrative Review. Mol Neurobiol. 2018 Aug;55(8):6601-6636. doi: 10.1007/s12035-017-0852-4. Epub 2018 Jan 11. PMID 29327206
- [Background] Tator CH. Concussions and their consequences: current diagnosis, management and prevention. CMAJ. 2013 Aug 6;185(11):975-9. doi: 10.1503/cmaj.120039. Epub 2013 Jul 22. No abstract available. PMID 23877672
- [Background] Zemek R, Barrowman N, Freedman SB, Gravel J, Gagnon I, McGahern C, Aglipay M, Sangha G, Boutis K, Beer D, Craig W, Burns E, Farion KJ, Mikrogianakis A, Barlow K, Dubrovsky AS, Meeuwisse W, Gioia G, Meehan WP 3rd, Beauchamp MH, Kamil Y, Grool AM, Hoshizaki B, Anderson P, Brooks BL, Yeates KO, Vassilyadi M, Klassen T, Keightley M, Richer L, DeMatteo C, Osmond MH; Pediatric Emergency Research Canada (PERC) Concussion Team. Clinical Risk Score for Persistent Postconcussion Symptoms Among Children With Acute Concussion in the ED. JAMA. 2016 Mar 8;315(10):1014-25. doi: 10.1001/jama.2016.1203. PMID 26954410
- [Background] Ruff RM. Mild traumatic brain injury and neural recovery: rethinking the debate. NeuroRehabilitation. 2011;28(3):167-80. doi: 10.3233/NRE-2011-0646. PMID 21558623
- See also: ICD 10 — https://icd.who.int/browse10/2019/en